CLINICAL TRIAL: NCT05262439
Title: Post Market Clinical Follow Up of ResMed Mask Systems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLP-21-12-01
Record Dates: First submitted 2022-02-03; First posted 2022-03-02 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- New generation CPAP mask (Experimental): The intended purpose of mask systems is to provide airflow from a CPAP device, through tubing, and to the patient. The air acts as a pneumatic splint to keep the airway open and prevent collapse during sleep. The masks to be used in this study are released masks approved and released.
  Interventions: Device: New generation CPAP mask

INTERVENTIONS:
Device: New generation CPAP mask — All participants entered into the study will be couriered a new generation ResMed mask system to be used with their own CPAP machine and in place of their own mask.

SUMMARY:
Post Market follow up study to systematically and proactively collect supplementary real world data to confirm the usability and performance of the new generation mask systems. .

DETAILED DESCRIPTION:
This is an open label, prospective, multi-centre, single arm study for post market clinical follow up. The study will be conducted in the home environment remotely. Eligible participants currently using older generations of CPAP masks will use the new generation ResMed mask system in the same mask category to their own (nasal, full face, pillow) in place of their own mask for 90 nights and complete a series of questionnaires at specified study checkpoints.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to give written informed consent
* Participants who can read and comprehend English
* Participants who ≥ 18 years of age
* Participants being treated for OSA for ≥ 6 months
* Participants currently using a suitable mask system
* Participants currently using CPAP device compatible with AirView, or with download capacity from CPAP machine from data cards

Exclusion Criteria:

* Participants using Bilevel flow generators
* Participants who are or may be pregnant
* Participants with a pre-existing lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury.
* Participants believed to be unsuitable for inclusion by the researcher
* Participants who or whose bed partner has implantable metallic implants in the head, neck and chest region affected by magnetic fields (Non-ferrous implants may be acceptable) (for masks with magnetic clips only)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (event/hour) | up to 90 days
  Apnea Hypopnea events per hour taken from the participant's CPAP device used during the study
Usage Hours (hours/night) | up to 90 days
  Average usage hours taken from the participant's CPAP device used during the study
Leak (L/minute) | up to 90 days
  Calculated leak from CPAP machine which assess how well mask seals on patients
CPAP Pressure (cmH2O) | up to 90 days
  Calculated average pressure from the CPAP machine which indicates how much pressure patients required to keep their airway open
Adverse Events | up to 90 days
  Device related adverse events during the study period will also be assessed.

SECONDARY OUTCOMES:
General Usability | up to 90 days
  Subjective usability scores from participants. Each usability item of the new mask system will be rated on a Likert Scale questionnaire. A score of 10 is considered very favourable whereas score of 0 is considered very unfavourable.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Armistead, PhD, Principal Investigator — ResMed
Locations (1):
- Medical Affairs ResMed, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu X, Benjafield A, Deas R, Willes L, Armitstead J. Feasibility and acceptability of switching from a previous-generation to a new-generation mask for positive airway pressure therapy of sleep apnea using remote care. Sleep Med X. 2024 Oct 11;8:100128. doi: 10.1016/j.sleepx.2024.100128. eCollection 2024 Dec 15. PMID 39498349